CLINICAL TRIAL: NCT07337967
Title: Reticulocyte Parameters as Early Indicators of Bone Marrow Erythropoietic Activity in Chronic B Lymphoproliferative Neoplasms
Status: Not yet recruiting | Type: Observational
Sponsor: Huda Ahmed Abdelsabour Abdelwahab (Other)
Responsible Party: Sponsor-Investigator, Huda Ahmed Abdelsabour Abdelwahab, Resident doctor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: AUN-FOM-CP-CLPD-RETIC-2025
Record Dates: First submitted 2025-12-13; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: B Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, B-Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Reticulocyte parameters as early indicators of bone marrow erythropoietic activity in chronic B lymphoproliferative neoplasms

ELIGIBILITY:
Inclusion Criteria:

- Newly diagnosed adult patients with Chronic B LymphoPoliferative neoplasm according to WHO classification.

Exclusion Criteria:

1) Patients received chemotherapy.

1. Patients with Active bleeding
2. Patients with recent blood transfusion (less than 2 weeks).
3. Patients on haematinics or vitamin B 12 therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed adult patients with Chronic B LymphoPoliferative neoplasm according to WHO classification.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Reticulocyte count | 1 year
  Absolute peripheral blood reticulocyte count measured in patients with chronic B-cell lymphoproliferative disorders (CLPDs).
  Unit of Measure: ×10⁹/L
Reticulocyte percentage | 1 year
  Percentage of reticulocytes among total red blood cells in peripheral blood of patients with CLPDs.
  Unit of Measure: %
Immature reticulocyte fraction (IRF) | 1 year
  Proportion of immature reticulocytes in peripheral blood measured in patients with CLPDs.
  Unit of Measure: %